CLINICAL TRIAL: NCT00391482
Title: Behavioral Intervention Trial to Reduce Transmission Risks and Improve HCV Treatment Access Among HCV-infected Injection Drug Users
Brief Title: Study to Reduce Intravenous Exposures (STRIVE)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DESPR DA014499; 1R01DA014499 (NIH)
Record Dates: First submitted 2006-10-20; First posted 2006-10-24 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2008-11

CONDITIONS: Hepatitis C; HIV Infections
Keywords: IV Drug Users; Hepatitis C Virus; Human Immunodeficiency Virus; Intervention; HIV Seronegativity
MeSH Terms: conditions — Hepatitis C; HIV Infections; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Behavioral: Peer Mentoring Intervention for HCV-Infected IDUs

SUMMARY:
The purpose of this study is to determine whether a six-session, small group behavioral intervention based on "peer-volunteer activism" is effective in (1) decreasing distributive sharing of syringes and other injection paraphernalia and (2) increasing utilization of HCV-related healthcare services among HCV-infected injection drug users

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy of a peer-volunteer intervention to reduce high-risk transmission behaviors among hepatitis C virus (HCV)-infected young adult injection drug users (IDUs), and to identify the proportion of these individuals who would be eligible and willing to undergo treatment to eradicate HCV infection. HCV is one of the most frequently occurring human viral infections, having an estimated worldwide prevalence of 3%. In many regions of the United States, between 65% and 95% of IDUs are HCV-seropositive and capable of transmitting the infection. To date, research studies targeting infected individuals to prevent secondary transmission of chronic blood-borne viral infection have generally been limited to post-test counseling and case management. In addition, recent data suggest that medical treatment of HCV infection may be most effective when offered soon after HCV seroconversion. However, the proportion of HCV-infected IDUs who meet strict national guidelines for HCV treatment is likely to be small because treatment is usually postponed while drug use continues. Determining the proportion of infected individuals who may be both eligible and willing to undergo HCV therapy is highly important for guiding national standards and objectives to achieve greater numbers of IDUs in HCV therapy. We have previously reported that fewer than 1% of HCV-infected IDUs in Baltimore are currently receiving such therapy. Early initiation of HCV treatment among young IDUs in conjunction with a reduction in HCV transmission risk behaviors may ultimately lead to a reduction in incident HCV infection at the individual and the community levels.

This study is a randomized controlled trial to determine the efficacy of a "peer-volunteer activism" intervention to reduce distributive syringe and injection paraphernalia sharing behaviors among HCV positive IDUs and promote the uptake of HCV care and treatment. If proven effective, this intervention would substantially decrease the risk of HCV infection in the community. To address these aims, we plan to recruit, screen, and randomly assign 750 IDUs age 18-35 years who are HCV-seropositive but HIV-seronegative in Baltimore, New York and Seattle to a behavioral intervention (250 per site), and prospectively monitor participants behavior at 3- and 6-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* HCV antibody positive
* age between 18 and 35 years old;
* reported injection drug use in the past 6 months
* willing to provide a blood sample for liver function testing

Exclusion Criteria:

* HIV antibody positive
* planned on moving from city within the next 12 months;
* unable to comprehend English well enough to complete English-only assessments and group sessions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 750
Dates: Start 2002-06; Study Completion 2005-02

PRIMARY OUTCOMES:
Self-reported frequency of distributive sharing of injection and non-injection drug equipment (i.e., lending, giving or selling used needles, syringes or paraphernalia to others)

SECONDARY OUTCOMES:
Alcohol use; disposal of syringes and paraphernalia; increased condom use; syringe exchange program use; readiness for HCV therapy and drug use cessation; and discussing HCV therapy options at a medical care visit.

CONTACTS AND LOCATIONS:
Overall Officials: Steffanie A Strathdee, PhD, Principal Investigator — Johns Hopkins University, Bloomberg School of Public Health,
Locations (3):
- United States (3):
  - Johns Hopkins University, Bloomberg School of Public Health, Baltimore, Maryland
  - New York Academy of Medicine, Center for Urban Epidemiologic Studies, New York, New York
  - Public Health Seattle & King County, Seattle, Washington

REFERENCES:
- [Background] Strathdee SA, Latka M, Campbell J, O'Driscoll PT, Golub ET, Kapadia F, Pollini RA, Garfein RS, Thomas DL, Hagan H; Study to Reduce Intravenous Exposures Project. Factors associated with interest in initiating treatment for hepatitis C Virus (HCV) infection among young HCV-infected injection drug users. Clin Infect Dis. 2005 Apr 15;40 Suppl 5(Suppl 5):S304-12. doi: 10.1086/427445. PMID 15768339
- [Background] Campbell JV, Hagan H, Latka MH, Garfein RS, Golub ET, Coady MH, Thomas DL, Strathdee SA; STRIVE Project. High prevalence of alcohol use among hepatitis C virus antibody positive injection drug users in three US cities. Drug Alcohol Depend. 2006 Feb 28;81(3):259-65. doi: 10.1016/j.drugalcdep.2005.07.005. Epub 2005 Aug 29. PMID 16129567
- [Background] Golub ET, Latka M, Hagan H, Havens JR, Hudson SM, Kapadia F, Campbell JV, Garfein RS, Thomas DL, Strathdee SA; STRIVE Project. Screening for depressive symptoms among HCV-infected injection drug users: examination of the utility of the CES-D and the Beck Depression Inventory. J Urban Health. 2004 Jun;81(2):278-90. doi: 10.1093/jurban/jth114. PMID 15136661
- [Background] Hagan H, Latka MH, Campbell JV, Golub ET, Garfein RS, Thomas DA, Kapadia F, Strathdee SA; Study to Reduce Intravenous Exposures Project Team. Eligibility for treatment of hepatitis C virus infection among young injection drug users in 3 US cities. Clin Infect Dis. 2006 Mar 1;42(5):669-72. doi: 10.1086/499951. Epub 2006 Jan 20. PMID 16447112
- [Derived] Drumright LN, Hagan H, Thomas DL, Latka MH, Golub ET, Garfein RS, Clapp JD, Campbell JV, Bonner S, Kapadia F, Thiel TK, Strathdee SA. Predictors and effects of alcohol use on liver function among young HCV-infected injection drug users in a behavioral intervention. J Hepatol. 2011 Jul;55(1):45-52. doi: 10.1016/j.jhep.2010.10.028. Epub 2010 Nov 24. PMID 21145862
- [Derived] Kapadia F, Latka MH, Hagan H, Golub ET, Campbell JV, Coady MH, Garfein RS, Thomas DL, Bonner S, Thiel T, Strathdee SA. Design and feasibility of a randomized behavioral intervention to reduce distributive injection risk and improve health-care access among hepatitis C virus positive injection drug users: the Study to Reduce Intravenous Exposures (STRIVE). J Urban Health. 2007 Jan;84(1):99-115. doi: 10.1007/s11524-006-9133-7. PMID 17200799